CLINICAL TRIAL: NCT03490929
Title: Contrast Enhanced Ultrasonography for Blunt Abdominal Trauma Imaging in Children
Brief Title: CEUS for Blunt Abdominal Trauma in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Aaron E. Chen, Professor of Clinical Pediatrics, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-014905
Record Dates: First submitted 2018-03-23; First posted 2018-04-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Trauma Abdomen
MeSH Terms: conditions — Abdominal Injuries | interventions — Suspensions; Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Contrast-enhanced ultrasound arm (Experimental): contrast-enhanced ultrasound
  Interventions: Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Intravenous Powder for Suspension [LUMASON]; Device: contrast-enhanced ultrasound

INTERVENTIONS:
Drug: Sulfur Hexafluoride Lipid Type A Microspheres 25 MG Intravenous Powder for Suspension [LUMASON] — injection of Lumason (ultrasound contrast agent)
  Other Names: Lumason
Device: contrast-enhanced ultrasound — ultrasound of the abdomen after injection of ultrasound contrast agent (Lumason)
  Other Names: ultrasound

SUMMARY:
Children with blunt abdominal trauma often get a CT as the first line imaging to evaluate for intra-abdominal organ injury. CT scans have some downsides with regard to radiation exposure, costs, and need for transport. Contrast enhanced ultrasonography has recently shown some promise as a way to detect intra-abdominal organ injury and may be able to replace the need for conventional CT scanning, without the need for ionizing radiation and the ability to be performed at the bedside.

DETAILED DESCRIPTION:
In children with abdominal trauma, computed tomography (CT) of the abdomen is considered the gold standard for the initial evaluation of solid organ injuries. The major drawbacks to CT include risks due to radiation exposure and necessity of transport of the patient. Ultrasound without contrast uses safer non-ionizing radiation and can be performed at the bedside, however it has been shown to have variable sensitivity and specificity for identifying intra-abdominal organ injury. Newer studies using contrast enhanced ultrasound (CEUS) have shown promise for improving the sensitivity and specificity of this imaging modality.

Hypothesis(es) and Aims:

Hypothesis: Contrast enhanced ultrasound (CEUS) has good sensitivity and specificity as compared to a gold standard conventional CT scan for the identification of intra-abdominal solid organ injury in hemodynamically stable children with blunt abdominal trauma. Specific Aims:

Primary Aim: To determine the test characteristics CEUS / conventional ultrasound for the detection of intra-abdominal solid organ injury, as compared to a gold standard CT scan, in hemodynamically stable children with blunt abdominal trauma

Design:

This will be a prospective cohort study to evaluate the test characteristics of contrast enhanced ultrasound (CEUS) for the detection of intra-abdominal solid organ injury in children with blunt abdominal trauma, as compared to a gold standard CT scan. Study subjects will be age 0-18 years, presenting with hemodynamically stable blunt abdominal trauma and for whom an abdominal CT scan is planned. The exclusion criteria will be a known allergy to the ultrasound contrast agent, co-existing penetrating abdominal trauma, or known congenital or acquired heart disease. Sample size calculations assume a baseline prevalence of disease in approximately 20% of patients receiving a CT scan, and target a sensitivity of at least 95% with a two-sided confidence interval precision of 8%, yielding an estimated sample size of 146 patients. The primary outcome will be calculation of sensitivity and specificity of CEUS as compared to a gold standard CT scan.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamically stable (defined as not needing massive transfusion protocol and not undergoing an emergent surgical procedure within the next hour)
2. History of or suspicion for blunt abdominal trauma
3. Abdominal CT ordered or obtained

Exclusion Criteria:

1. History of allergic reaction to Lumason, sulfur hexaflouride, sulfur hexafluoride lipid microsphere components, or other ingredients in Lumason (polyethylene glycol, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), palmitic acid)
2. Co-existing penetrating abdominal trauma
3. Known congenital or acquired heart disease

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of CEUS | through study completion, which is expected to take around 3 years
  calculation of sensitivity of CEUS for organ injury, as compared to gold standard CT
Specificity of CEUS | through study completion, which is expected to take around 3 years
  calculation of specificity of CEUS for organ injury, as compared to gold standard CT exam

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Chen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Armstrong LB, Mooney DP, Paltiel H, Barnewolt C, Dionigi B, Arbuthnot M, Onwubiko C, Connolly SA, Jarrett DY, Zalieckas JM. Contrast enhanced ultrasound for the evaluation of blunt pediatric abdominal trauma. J Pediatr Surg. 2018 Mar;53(3):548-552. doi: 10.1016/j.jpedsurg.2017.03.042. Epub 2017 Mar 20. PMID 28351519
- [Background] Miele V, Piccolo CL, Galluzzo M, Ianniello S, Sessa B, Trinci M. Contrast-enhanced ultrasound (CEUS) in blunt abdominal trauma. Br J Radiol. 2016;89(1061):20150823. doi: 10.1259/bjr.20150823. Epub 2016 Jan 8. PMID 26607647
- [Background] Menichini G, Sessa B, Trinci M, Galluzzo M, Miele V. Accuracy of contrast-enhanced ultrasound (CEUS) in the identification and characterization of traumatic solid organ lesions in children: a retrospective comparison with baseline US and CE-MDCT. Radiol Med. 2015 Nov;120(11):989-1001. doi: 10.1007/s11547-015-0535-z. Epub 2015 Mar 31. PMID 25822953
- [Background] Cagini L, Gravante S, Malaspina CM, Cesarano E, Giganti M, Rebonato A, Fonio P, Scialpi M. Contrast enhanced ultrasound (CEUS) in blunt abdominal trauma. Crit Ultrasound J. 2013 Jul 15;5 Suppl 1(Suppl 1):S9. doi: 10.1186/2036-7902-5-S1-S9. Epub 2013 Jul 15. PMID 23902930
- [Background] Cokkinos D, Antypa E, Stefanidis K, Tserotas P, Kostaras V, Parlamenti A, Tavernaraki K, Piperopoulos PN. Contrast-enhanced ultrasound for imaging blunt abdominal trauma - indications, description of the technique and imaging review. Ultraschall Med. 2012 Feb;33(1):60-7. doi: 10.1055/s-0031-1273442. Epub 2012 Jan 24. PMID 22274907
- [Background] Afaq A, Harvey C, Aldin Z, Leen E, Cosgrove D. Contrast-enhanced ultrasound in abdominal trauma. Eur J Emerg Med. 2012 Jun;19(3):140-5. doi: 10.1097/MEJ.0b013e328348c980. PMID 21934507
- [Background] Valentino M, De Luca C, Galloni SS, Branchini M, Modolon C, Pavlica P, Barozzi L. Contrast-enhanced US evaluation in patients with blunt abdominal trauma(). J Ultrasound. 2010 Mar;13(1):22-7. doi: 10.1016/j.jus.2010.06.002. Epub 2010 Jul 8. PMID 23396012
- [Background] Valentino M, Ansaloni L, Catena F, Pavlica P, Pinna AD, Barozzi L. Contrast-enhanced ultrasonography in blunt abdominal trauma: considerations after 5 years of experience. Radiol Med. 2009 Oct;114(7):1080-93. doi: 10.1007/s11547-009-0444-0. Epub 2009 Sep 22. PMID 19774445
- [Background] Sivit CJ. Imaging children with abdominal trauma. AJR Am J Roentgenol. 2009 May;192(5):1179-89. doi: 10.2214/AJR.08.2163. PMID 19380540
- [Background] Catalano O, Aiani L, Barozzi L, Bokor D, De Marchi A, Faletti C, Maggioni F, Montanari N, Orlandi PE, Siani A, Sidhu PS, Thompson PK, Valentino M, Ziosi A, Martegani A. CEUS in abdominal trauma: multi-center study. Abdom Imaging. 2009 Mar-Apr;34(2):225-34. doi: 10.1007/s00261-008-9452-0. PMID 18682877
- [Background] Clevert DA, Weckbach S, Minaifar N, Clevert DA, Stickel M, Reiser M. Contrast-enhanced ultrasound versus MS-CT in blunt abdominal trauma. Clin Hemorheol Microcirc. 2008;39(1-4):155-69. PMID 18503121
- [Background] Valentino M, Serra C, Pavlica P, Labate AM, Lima M, Baroncini S, Barozzi L. Blunt abdominal trauma: diagnostic performance of contrast-enhanced US in children--initial experience. Radiology. 2008 Mar;246(3):903-9. doi: 10.1148/radiol.2463070652. Epub 2008 Jan 14. PMID 18195385
- [Background] Bixby SD, Callahan MJ, Taylor GA. Imaging in pediatric blunt abdominal trauma. Semin Roentgenol. 2008 Jan;43(1):72-82. doi: 10.1053/j.ro.2007.08.009. No abstract available. PMID 18053830
- [Background] Ntoulia A, Anupindi SA, Darge K, Back SJ. Applications of contrast-enhanced ultrasound in the pediatric abdomen. Abdom Radiol (NY). 2018 Apr;43(4):948-959. doi: 10.1007/s00261-017-1315-0. PMID 28980061
- [Background] Darge K, Papadopoulou F, Ntoulia A, Bulas DI, Coley BD, Fordham LA, Paltiel HJ, McCarville B, Volberg FM, Cosgrove DO, Goldberg BB, Wilson SR, Feinstein SB. Safety of contrast-enhanced ultrasound in children for non-cardiac applications: a review by the Society for Pediatric Radiology (SPR) and the International Contrast Ultrasound Society (ICUS). Pediatr Radiol. 2013 Sep;43(9):1063-73. doi: 10.1007/s00247-013-2746-6. Epub 2013 Jul 11. PMID 23843130
- [Background] Parker JM, Weller MW, Feinstein LM, Adams RJ, Main ML, Grayburn PA, Cosgrove DO, Goldberg BA, Darge K, Nihoyannopoulos P, Wilson S, Monaghan M, Piscaglia F, Fowlkes B, Mathias W, Moriyasu F, Chammas MC, Greenbaum L, Feinstein SB. Safety of ultrasound contrast agents in patients with known or suspected cardiac shunts. Am J Cardiol. 2013 Oct 1;112(7):1039-45. doi: 10.1016/j.amjcard.2013.05.042. Epub 2013 Jun 28. PMID 23816393